CLINICAL TRIAL: NCT01126372
Title: Prediction of Feeding Problems in Prostaglandin-dependent Prematurely Born Infants With Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Christian Con Yost, University of Utah
Other Study IDs: 40795
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Congenital Heart Disease; Prematurity; Necrotizing Enterocolitis
Keywords: Prostaglandin-dependent Congenital Heart Disease; Prematurity; Feeding intolerances; Necrotizing Enterocolitis; Regional Oxygen Saturation; Near Infrared Spectroscopy; Somanetics INVOS Oxyalert
MeSH Terms: conditions — Heart Defects, Congenital; Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Prematurely born infants with ductal-dependent congenital heart disease (CHD) are at increased risk to develop necrotizing enterocolitis (NEC). Abnormal left to right blood flow through a patent ductus arteriosus can cause intestinal ischemia and compromise the gastrointestinal tract as a barrier to infection. In some infants, bacterial translocation leads to NEC which may result in death, intestinal perforation, cholestasis and, at the very least, feeding problems. Predicting which infants with CHD will develop NEC will potentially decrease the severity of disease if interventions were started earlier.

Near-infrared spectroscopy (NIRS) allows determination of regional oxygen saturation levels in tissues such as brain, kidney, and as recently reported, intestine. This study will test whether or not decreasing intestinal oxygen saturations can predict the development of NEC in this at risk population before the symptoms become severe. NIRS probes will be placed on the forehead, flank and abdomen of eligible infants and regional oxygen saturations will be recorded prospectively and continuously with the clinical care team blinded to the data. The development of NEC and significant feeding problems will then be correlated with the regional oxygen saturations to determine whether decreased intestinal oxygen saturations predicted early signs and symptoms of NEC.

We anticipate generating pilot data in 30 infants who meet inclusion criteria. Support of this research will be provided partially by Somanetics, the manufacturer of the INVOS regional oxygen saturation monitors. They will, however, have no control over the data generated by this study.

ELIGIBILITY:
Inclusion Criteria:

* >/+ 30 and 0/7 weeks gestation age at birth
* Anticipated time to surgical repair is > 7 days
* Meets criteria for management via the PCMC CHD feeding protocol

Exclusion Criteria:

* Any extracardiac major congenital anomalies

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted into the NICU at PCMC (Salt Lake City, UT) with a prostaglandin-dependent congenital heart defect (CHD).
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Evaluate intestinal oxygen saturations using NIRS to predict the development of NEC. | 2 months
  Using NIRS to test whether or not decreasing intestinal oxygen saturations can predict the development of NEC in this at risk population before the symptoms become severe.

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Yost, MD, Principal Investigator — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States